CLINICAL TRIAL: NCT03587155
Title: Study on the Mechanism of Neurodevelopment Dysplasia of Fetal Brain Caused by ASNS Gene Mutation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Bo Chen, Associate Chief Physician, The First Hospital of Jilin University
Other Study IDs: ASNS-BRAIN001
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Asparagine Synthetase Deficiency; Genetic Diseases, Inborn
Keywords: ASNS, single cell RNA seq, Neurodevelopmental Dysplasia,
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extract DNA from brain tissue or peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mutation: Embryo or infant with ASNS mutation.
- Control: Embryo or infant without ASNS mutation.

SUMMARY:
The investigators propose to analyze a brain sample and/or peripheral blood by single cell RNA seq from aborted embryos with ASNS mutation.

DETAILED DESCRIPTION:
Congenital microcephaly could cause by gene mutation. Asparagine synthetase deficiency, which is caused by ASNS mutation, is a rare autosomal recessive neurometabolic disorder. It is characterized by severe developmental delay, congenital microcephaly, seizures. The investigators found a family with ASNS mutaion. The investigators propose to analyze a brain sample and/or peripheral blood by single cell RNA seq from aborted embryos with ASNS mutation.

ELIGIBILITY:
Inclusion Criteria:

* Mutation Group: Having ASNS gene mutation by DNA exon sequencing.
* Control Group: No ASNS gene mutation by DNA exon sequencing.

Exclusion Criteria:

* Mutation Group: N/A.
* Control Group: Having other gene mutation which also effect neurodevelopment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: abortive embryo or infant.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Effect of ASNS gene mutation on RNA expression in prefrontal cortex cells of brain tissue | 2018.06-2020.12
  Detect RNA expression in prefrontal cortex cells by single cell RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Chen, M.D., Ph.D., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Bo Chen, Changchun, Jilin, China